CLINICAL TRIAL: NCT01398267
Title: A Randomized, Double-blind, Placebo-controlled, Parallel Group Study to Investigate the Effects of Aleglitazar 150 µg in Type 2 Diabetic Patients Treated With Lisinopril 20 mg on Renal Function, the Renin-angiotensin System and the Pharmacokinetics of Lisinopril
Brief Title: A Pharmacodynamic/Pharmacokinetic Study of Aleglitazar in Patients With Type 2 Diabetes Mellitus on Treatment With Lisinopril
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double
Other Study IDs: BP25328
Record Dates: First submitted 2011-07-19; First posted 2011-07-20 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Diabetes Mellitus Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — aleglitazar; Lisinopril

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- 1 (Experimental)
  Interventions: Drug: aleglitazar; Drug: lisinopril
- 2 (Placebo Comparator)
  Interventions: Drug: lisinopril; Drug: placebo

INTERVENTIONS:
Drug: aleglitazar — 150 mcg orally daily, 4 weeks (Day 15 to Day 43)
  Arms: 1
Drug: lisinopril — 20 mg orally daily, 6 weeks (Day 1 to Day 43)
Drug: placebo — aleglitazar matching placebo orally daily, 4 weeks (Day 15 to Day 43)
  Arms: 2

SUMMARY:
This randomized, double-blind, placebo-controlled, parallel-group study will evaluate the effect of aleglitazar on renal function, the renin-angiotensin system and the pharmacokinetics of lisinopril in patients with type 2 diabetes mellitus treated with lisinopril. Patients on a stable dose of lisinopril (20 mg daily orally) for 2 weeks will be randomized to receive either aleglitazar (150 mcg orally daily) or placebo in addition to lisinopril for 4 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Adult male and female patients, 18 to 65 years of age, inclusive
* Diabetes mellitus Type 2, diagnosed at least 3 months before screening
* Treated with stable dose of metformin for at least 4 weeks prior to screening
* Treated with stable dose of Angiotensin-converting enzyme inhibitor (ACEI) for at least 4 weeks prior to screening
* Body mass index (BMI) 18 to 38 kg/m2, inclusive

Exclusion Criteria:

* Positive for HIV-1, HIV-2, hepatitis B or hepatitis C infection
* Pregnant or lactating females
* Type 1 diabetes or secondary from of diabetes
* History or evidence of proliferative diabetic retinopathy or clinically significant neuropathy
* Clinically significant hepatic disease
* Clinically significant renal impairment
* History or evidence of clinically significant cardio-vascular disease or disorder
* Acute infection or current malignancy requiring treatment except for excised basal cell carcinoma

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2011-08; Primary Completion 2012-10 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Glomerular filtration rate (mGFR), measured as iohexol clearance | 4 weeks

SECONDARY OUTCOMES:
Estimated glomerular filtration rate, using modification of diet in renal disease formula (eGFR[MDRD]) | 4 weeks
Effective renal plasma flow rate (ERPF), measured as Para-amino hippuric acid (PAH) clearance (PAH plasma concentrations) | 4 weeks
Electrolyte blood/urine concentrations | 4 weeks
Renin-angiotensin system: plasma renin/aldosterone levels) | 4 weeks
Anti-diuretic hormone (ADH) blood levels | 4 weeks
Safety: Incidence of adverse events | up to 18 weeks
Effect of multiple doses of aleglitazar on lisinopril steady-state pharmacokinetics (area under the concentration - time curve [AUC]) | 4 weeks
Steady-state pharmacokinetics (AUC) of aleglitazar in co-administration with lisinopril | 4 weeks
High density lipoprotein-cholesterol (HDL-C) blood levels | 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (4):
- United States (4):
  - Chula Vista, California
  - Omaha, Nebraska
  - Dallas, Texas
  - San Antonio, Texas